CLINICAL TRIAL: NCT05853679
Title: Effect of Regular Antibacterial Photodynamic Therapy on Oral Hygiene in Elderly Residents of a 24-hour Care Facility
Brief Title: Regular Antibacterial Photodynamic Therapy on Oral Hygiene in Elderly Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: University of Helsinki (Other); City of Helsinki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSAA2021
Record Dates: First submitted 2023-04-21; First posted 2023-05-11 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Dental Plaque; Pus Collection; Oral Disease; Dryness Oral; Tooth Decay
Keywords: Lumoral; Lumorinse; Plaque Control; Anti-bacterial photodynamic therapy; aMMP-8; Care home
MeSH Terms: conditions — Dental Plaque; Mouth Diseases; Xerostomia; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization of patients is done by using sealed envelope technique at the end of the Baseline visit. During the Baseline visit, participants, care providers, and investigators do not know to which group the participant will be allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumoral Treatment (Study group) (Experimental): A complete clinical intraoral examination shall be performed for all subjects. Same demographic and clinical data will be obtained from subjects in both arms. The study group shall receive the Lumoral treatment -device, Lumorinse -tablets and instructions for their use.
  All subjects shall receive new electric toothbrushes, standard oral hygiene instructions for the use of an electric toothbrush, interdental brush, and dental floss.
  Interventions: Device: Lumoral Treatment
- Control group (Other): A complete clinical intraoral examination shall be performed for all subjects. Same demographic and clinical data will be obtained from subjects in both arms. All subjects shall receive new electric toothbrushes, standard oral hygiene instructions for the use of an electric toothbrush, interdental brush, and dental floss.
  Interventions: Device: Lumoral Treatment; Other: Standard oral hygiene instructions according to the Finnish Dental Association

INTERVENTIONS:
Device: Lumoral Treatment — The device will be used 5 to 7 times per week according to the manufacturer's instructions.
Other: Standard oral hygiene instructions according to the Finnish Dental Association — Participants will be instructed to clean their teeth twice per day by an electric toothbrush, an interdental brush, and flossing.
  Arms: Control group

SUMMARY:
Around 40 people will participate in the study. The study participants will be recruited from service homes in the City of Helsinki. The subjects will be randomized into two groups. One of the groups will receive daily photodynamic Lumoral treatment for 2 months in a home care unit according to a separate instruction manual. At the beginning of the study, all subjects will receive an oral cleaning and will also be provided with electric toothbrushes. In addition, residents and care home personnel will be instructed on daily tooth cleaning.

During the study, all participants will undergo clinical measurements and an assessment of the oral inflammatory load. The samples will be stored for later analysis. In addition, residents or care home personnel answer questions about oral self-care. These measurements and examinations will be carried out at the start of the study and two months after the start of the study. After the end of the study, participants will continue to be treated according to their usual care and individual care plan.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of regular antibacterial photodynamic treatment in service accommodation on the oral hygiene of elderly people. The information from this study can be used to promote oral hygiene among residents in 24-hour care.

Lumoral is a CE-marked medical home appliance that has been shown to be effective in reducing plaque development and the amount of harmful bacteria in plaque. The efficacy of the device is based on an antibacterial photodynamic process, whereby a photosensitive substance in Lumorinse attaches itself to the bacterial coating and is activated as an antibacterial agent by light. The antibacterial effect is directly targeted at the plaque, reducing the impact on the normal oral flora. Preliminary studies have shown that the method reduces the inflammatory factors associated with periodontitis.

The study is being carried out in collaboration with the City of Helsinki Oral Health Department, the Metropolia University of Applied Sciences Oral Care Teaching Hospital and the University of Helsinki Department of Oral and Maxillofacial Surgery. The registrar of the study is the University of Helsinki. The study will be conducted in accordance with Good Clinical Practice (GCP) and ISO 14155 ("Clinical trials on medical devices. Good Clinical Practice").

The target population of the study will be residents in 24-hour care with at least 10 of their own teeth, who are judged by the caregiver to be able to participate in the study and who give written informed consent to participate in the study.

Approximately 40 people will participate in the study. They will be recruited from the City of Helsinki's service homes. The subjects will be randomized into two groups. One of the groups will receive daily photodynamic Lumoral treatment for 2 months in a residential unit according to a separate instruction manual. At the beginning of the study, all subjects will receive an oral cleaning and will also be provided with electric toothbrushes. In addition, residents and carers will be instructed on daily tooth cleaning.

During the study, all patients will undergo clinical measurements (VPI, CPITN, dry mouth) and an assessment of the oral inflammatory load using the aMMP-8 bowel inflammation test. The occlusion samples will be stored for later analysis. In addition, residents or caregivers answer questions about oral self-care. These measurements and examinations will be carried out at the start of the study and two months after the start of the study. After the end of the study, subjects will continue to be treated according to their usual care and individual care plan.

ELIGIBILITY:
Inclusion Criteria:

* A 24-hour care resident;
* Understand and able to give consent to the study;
* At least 10 functional teeth in the mouth (including implants);
* Able to brush teeth and follow the instruction for use Lumoral treatment, based on the assessment by the nursing staff.

Exclusion Criteria:

* Incapable of participating in the study based on the assessment of the nursing staff
* Toothless or less than 10 functional teeth in the mouth (including implants)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Change in oral hygiene / patient experience | 2 months
  A change in baseline oral self-care and hygiene questionnaire compared to 2-month follow-up.
  The questionnaires are completed by the study participants.
Visible Plaque Index | 2 months
  Change in Visible Plaque Index:
  * A full-mouth assessment at 4 sites per tooth will be made at baseline and at the 2 month follow-up visit
  * VPI is reported as the percentage (%) of sites with positive findings
  * Dichotomous scoring to each site of the tooth as plaque" 1 present" and" 0 absent"
  * Calculation formula: number of plaque sites/ 4 times number of teeth
aMMP-8 chaiside test | 2 months
  Change in oral inflammatory load measured by the aMMP-8 chairside speed test:
  * The aMMP-8 marker analysis will be performed using the Periosafe chair-side test (Dentognostics GmbH) according to the manufacturer's instructions.
  * Oral rinse samples will be stored for further analysis.
  * Further analysis includes aMMP-8 and its regulators by biochemical enzyme/molecule assays, immunoassays, and proteomics analysis.

SECONDARY OUTCOMES:
Dryness in mouth | 2 months
  Change in dryness in mouth. The data will be obtained by the thorough oral inspection performed by the investigators, and by a questionnaire (patient outcome).
  Clinical assessment of moisture/dryness of oral mucosa (score 0-2):
  0 = Saliva secretion looks normal (saliva serous and running)
  1. = Mucous membrane of the mouth shiny and tightening/ saliva foamy or mucous/ little clear saliva at the base of the mouth
  2. = Mouth completely dry, mirror sticking to cheek or tongue, mucous membranes often reddened/ bumps on tongue surface disappeared/ scab on melting.
Dryness in mouth (patient experience) | 2 months
  The data will be obtained by a oral health questionnaire (patient outcome).
Usability of Lumoral Treatment device (patient outcome) | 2 months
  The study participants will answer a questionnaire related to the usability of Lumoral Treatment device.
Usability of Lumoral Treatment device (care home personnel outcome) | 2 months
  The care home nursing staff will answer a questionnaire related to their view of the usability of Lumoral Treatment device. The questionnaire will also ask about how easy or hard it was to instruct the care home patients to use the device on a near-daily basis and if they would recommend the device for further use or to their customers.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Sorsa, Professor, Principal Investigator — University of Helsinki; Riitta Saarela, Study Chair — City of Helsinki; Tommi Pätilä, Study Director — Helsinki University Central Hospital
Locations (1):
- City of Helsinki, Health and Social Services, Senior Services, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Visschere L, de Baat C, De Meyer L, van der Putten GJ, Peeters B, Soderfelt B, Vanobbergen J. The integration of oral health care into day-to-day care in nursing homes: a qualitative study. Gerodontology. 2015 Jun;32(2):115-22. doi: 10.1111/ger.12062. Epub 2013 Jun 20. PMID 23786637
- [Background] Lahteenmaki H, Patila T, Raisanen IT, Kankuri E, Tervahartiala T, Sorsa T. Repeated Home-Applied Dual-Light Antibacterial Photodynamic Therapy Can Reduce Plaque Burden, Inflammation, and aMMP-8 in Peri-Implant Disease-A Pilot Study. Curr Issues Mol Biol. 2022 Mar 8;44(3):1273-1283. doi: 10.3390/cimb44030085. PMID 35723308
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Nothdurft HD, Jelinek T, Pechel SM, Hess F, Maiwald H, Marschang A, von Sonnenburg F, Weinke T, Loscher T. Stand-by treatment of suspected malaria in travellers. Trop Med Parasitol. 1995 Sep;46(3):161-3. PMID 8533018
- [Background] Nishizawa T, Niikura Y, Akasaka K, Watanabe M, Kurai D, Amano M, Ishii H, Matsushima H, Yamashita N, Takizawa H. Pilot study for risk assessment of aspiration pneumonia based on oral bacteria levels and serum biomarkers. BMC Infect Dis. 2019 Sep 2;19(1):761. doi: 10.1186/s12879-019-4327-2. PMID 31477059
- [Background] Saarela RKT, Hiltunen K, Mantyla P, Pitkala KH. Changes in Institutionalized Older People's Dentition Status in Helsinki, 2003-2017. J Am Geriatr Soc. 2020 Jan;68(1):221-223. doi: 10.1111/jgs.16230. Epub 2019 Oct 26. No abstract available. PMID 31654530
- [Background] Saarela RKT, Hiltunen K, Kautiainen H, Roitto HM, Mantyla P, Pitkala KH. Oral hygiene and health-related quality of life in institutionalized older people. Eur Geriatr Med. 2022 Feb;13(1):213-220. doi: 10.1007/s41999-021-00547-8. Epub 2021 Jul 27. PMID 34313976
- [Background] Suominen AL, Varsio S, Helminen S, Nordblad A, Lahti S, Knuuttila M. Dental and periodontal health in Finnish adults in 2000 and 2011. Acta Odontol Scand. 2018 Jul;76(5):305-313. doi: 10.1080/00016357.2018.1451653. Epub 2018 Mar 16. PMID 29546776
- [Background] Willumsen T, Karlsen L, Naess R, Bjorntvedt S. Are the barriers to good oral hygiene in nursing homes within the nurses or the patients? Gerodontology. 2012 Jun;29(2):e748-55. doi: 10.1111/j.1741-2358.2011.00554.x. Epub 2011 Oct 24. PMID 22023222
- See also: Hiltunen K, Julkunen L, Vesa T et al. 2020. Residents' oral health in long-term 24-hour care for the elderly in Helsinki 2018, Studies and reports of the Social and Health Services Department, City of Helsinki Social and Health Services Department — https://www.hel.fi/static/sote/julkaisut/asukkaiden-suunterveys-iakkaiden-pitkaaikaisessa-ymparivuorokautisessa-hoidossa.pdf
- See also: Suominen L, Vehkalahti M, Knuutila M. Health, functional capacity and well-being in Finland 2011. THL report 68/2012. — https://www.julkari.fi/bitstream/handle/10024/90832/Rap068_2012_netti.pdf?sequence=1&isAllowed=y